CLINICAL TRIAL: NCT06728228
Title: Amnioinfusion for Fetal Renal Failure
Status: Recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: Fetal Care Center, PLLC (Industry)
Collaborators: Medical City Children's Hospital (Other); Medical City Women's Hospital (Unknown)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: 2063654
Record Dates: First submitted 2024-12-06; First posted 2024-12-11 (Actual); Last update posted 2024-12-20 (Actual); Status verified 2024-12

CONDITIONS: Multicystic Dysplastic Kidney; Polycystic Kidney Disease; Fetal Renal Anomaly; Anhydramnios; Potter Syndrome; Lung Hypoplasia; Multicystic Renal Dysplasia, Bilateral; Lower Urinary Tract Obstructive Syndrome; Bilateral Renal Agenesis
Keywords: Fetal Renal Failure; Kidney Disease; MCDK; PCKD
MeSH Terms: conditions — Multicystic Dysplastic Kidney; Polycystic Kidney Diseases; Hereditary renal agenesis; Multicystic renal dysplasia, bilateral; Kidney Diseases

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (2):
- Amnioinfusion (Experimental): Those in this experimental arm, Amnioinfusion, will undergo serial amnioinfusion in addition to routine care as deemed appropriate by the study doctor.
  Interventions: Other: Amnioinfusion
- Comfort Care/Expectant Management (No Intervention): The non-experimental arm, Comfort Care/Expectant Management, will undergo comfort care as elected by the participant.

INTERVENTIONS:
Other: Amnioinfusion — A 20- or 22-gauge spinal needle (routinely used obstetrics and gynecology needle) will be used by an expert in fetal procedures with sterile technique to access the amniotic cavity under real-time ultrasound guidance to infuse isotonic fluid (Lactated Ringers with 1g/L of Oxacillin). This fluid will act as replacement amniotic fluid. Regular monitoring of fluid levels may suggest serial infusion, which will be completed as deemed necessary by the study doctor.
  Other Names: Amniotic fluid injection
  Arms: Amnioinfusion

SUMMARY:
The goal of this clinical trial is to learn if serial amnioinfusions can improve the chances of survival for fetuses with severe kidney problems that cause low amniotic fluid (anhydramnios). Low amniotic fluid can affect lung development and may lead to serious health issues for the fetus. The main questions this study aims to answer are:

* Can serial amnioinfusion increase the chances of survival for these fetuses?
* Does this procedure improve chances of survival until dialysis and/or kidney transplant?

Participants will:

* Receive regular amnioinfusions, which is a procedure that adds fluid to the amniotic cavity.
* Undergo monitoring to check the effects on the fetus and mother.

This study will help researchers understand if amnioinfusion is a useful treatment for fetal kidney problems and may provide valuable information for similar cases in the future.

DETAILED DESCRIPTION:
Fetal renal failure (FRF) is a severe and life-threatening condition caused by congenital abnormalities or inherited kidney diseases. In the womb, when the kidneys fail to function properly, this leads to a condition called anhydramnios-a complete lack of amniotic fluid. Amniotic fluid is essential for the fetus's lung development, particularly during the canalicular phase of pulmonary development, which occurs between 16 and 28 weeks of gestation. Without sufficient amniotic fluid, the lungs cannot develop properly, resulting in a condition known as pulmonary hypoplasia. Severe hypoplasia has previously been described as almost always fatal, typically leading to neonatal death shortly after birth.

In recent years, promising advances in fetal therapies have opened new doors for treating conditions that were once considered untreatable. One such intervention involves serial amnioinfusion, a procedure where sterile saline or another isotonic fluid is injected into the amniotic sac to restore fluid levels. Early studies, including the RAFT trial (Renal Anhydramnios Fetal Therapy), have demonstrated that this approach may improve survival rates by promoting lung development in fetuses with FRF. Building upon these findings, this study seeks to further evaluate the safety and effectiveness of serial amnioinfusion in improving neonatal outcomes for families facing this diagnosis.

This study will enroll approximately 60 pregnant individuals carrying singleton pregnancies complicated by FRF and anhydramnios. Participants will be divided into two groups: an intervention group, which will receive serial amnioinfusion procedures as deemed appropriate by the study doctor, and a control group, which will not undergo interventions and will receive comfort care for their pregnancies. The primary goals of the study are to evaluate maternal safety, assess fetal survival to dialysis, and determine survival to kidney transplant eligibility.

The amnioinfusion procedures will be performed at the Fetal Care Center by a team of experts in fetal procedures. To ensure patient safety, the study includes a rigorous monitoring plan to track any potential adverse events in real time. Data from imaging studies (e.g., ultrasound, echocardiogram, MRI) and laboratory biomarkers will be collected to evaluate fetal and maternal responses to the treatment. While the study focuses on improving outcomes for individual patients, it also has broader implications for science and society. By systematically analyzing the benefits and risks of serial amnioinfusion, this research could help refine treatment protocols and set the stage for new standards of care for FRF. For the families involved, participation in this study offers the possibility of improved survival for their children, with potential eligibility for life-saving kidney transplants in the future.

This study represents a critical step toward addressing a condition that has long been considered untreatable. Through collaboration, innovation, and rigorous research, the team aims to provide hope for families affected by FRF.

ELIGIBILITY:
Inclusion criteria:

1. Confirmed anhydramnios before 22 weeks GA for patients with FRF.
2. Consent is signed and first therapeutic amnioinfusion can and does occur before 28 weeks and 6/7 days GA.
3. Confirmation that the expectant mother understands her options for management of the pregnancy.
4. Age ≥18 years of age.
5. Willingness to be followed by the Fetal Care Center at Dallas and deliver at Medical City Dallas.
6. Willingness for postnatal care to be performed at Medical City Dallas Hospital/the Fetal Care Center until maternal discharge.
7. Consults with Pediatric Nephrology, Neonatology, Transplant Surgery, Pediatric surgery, Maternal-Fetal Medicine Specialist, and a Genetic Counselor.

Exclusion criteria:

1. Cervix less than 2.5 cm in length.
2. No fatal findings on Karyotype (e.g trisomy 13, or 18) or Microarray fatal findings excluding those that are related to pulmonary hypoplasia due to fetal renal failure (e.g. Meckel-Gruber, PCKD).
3. Other significant congenital anomalies in the fetus.
4. Evidence of chorioamnionitis or abruptio placentae.
5. Evidence of rupture of membranes or chorionic-amniotic separation.
6. Evidence of preterm labor.
7. Multiple gestation.
8. Severe maternal medical condition in pregnancy.
9. Clinically diagnosed maternal depression, psychoses, or anxiety that are refractory to treatment.
10. Technical limitations precluding amnioinfusion.

Sex: Female | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Gender Based: Yes — This study only accepts pregnant women.
Enrollment: 35 (Estimated)
Dates: Start 2024-12-05 (Actual); Primary Completion 2025-11-15 (Estimated); Study Completion 2026-11-15 (Estimated)

PRIMARY OUTCOMES:
Fetal Survival to Dialysis | Birth to either survival to >=14 days and placement of dialysis access, or nonsurvival, up to 3 weeks.
  Proportion of neonates surviving to >= 14 days and placement of dialysis access after serial amnioinfusions (defined as use of a dialysis catheter for >=14 continuous days)
Fetal Survival to Transplant | >=2 years after delivery.
  The proportion of neonates who survive to receive a kidney transplant following continuous, successful dialysis.
Incidence of Maternal Treatment-Emergent Adverse Events [Safety and Tolerability] | From enrollment in the study through delivery and up to 30 days postpartum.
  Maternal safety will be assessed by tracking adverse events, including bleeding, infections, and preterm rupture of membranes, at each visit, after procedures, and postpartum. These events will be documented at each prenatal visit, following every amnioinfusion, at delivery, and during a follow-up period of at least 30 days postpartum. The safety evaluation will focus on identifying procedure-related complications and ensuring the well-being of participants throughout the study.

SECONDARY OUTCOMES:
Number of infusions prior to rupture of membranes among participants in the intervention group | During the pregnancy, up to 9 months
  The practicality of performing serial amnioinfusions for early pregnancy renal anhydramnios will be evaluated by counting the number of infusions administered before rupture of membranes in the intervention group.
Mean gestational age at rupture of membranes in the intervention group | During the pregnancy, up to 9 months
  The feasibility of serial amnioinfusions will be assessed by determining the average gestational age at which rupture of membranes occurs in the intervention group.
Mean gestational age at delivery in the intervention group | During the pregnancy, up to 9 months
  The feasibility of serial amnioinfusions will be measured by calculating the mean gestational age at delivery among participants in the intervention group.
Rate of fetal demise in utero among participants in the non-intervention group | During the pregnancy, up to 9 months
  An exploratory analysis will examine the natural progression of untreated early pregnancy renal anhydramnios by analyzing the rate of in utero fetal demise in the non-intervention group.
Mean gestational age at delivery in the non-intervention group | During the pregnancy, up to 9 months
  An exploratory study will investigate the natural history of untreated early pregnancy renal anhydramnios by calculating the average gestational age at delivery for participants in the non-intervention group.

CONTACTS AND LOCATIONS:
Locations (1):
- Fetal Care Center, Dallas, Texas, United States

IPD SHARING:
Plan to Share IPD: Undecided

REFERENCES:
- [Background] Miller JL, Baschat AA, Rosner M, Blumenfeld YJ, Moldenhauer JS, Johnson A, Schenone MH, Zaretsky MV, Chmait RH, Gonzalez JM, Miller RS, Moon-Grady AJ, Bendel-Stenzel E, Keiser AM, Avadhani R, Jelin AC, Davis JM, Warren DS, Hanley DF, Watkins JA, Samuels J, Sugarman J, Atkinson MA. Neonatal Survival After Serial Amnioinfusions for Bilateral Renal Agenesis: The Renal Anhydramnios Fetal Therapy Trial. JAMA. 2023 Dec 5;330(21):2096-2105. doi: 10.1001/jama.2023.21153. PMID 38051327
- [Background] O'Hare EM, Jelin AC, Miller JL, Ruano R, Atkinson MA, Baschat AA, Jelin EB. Amnioinfusions to Treat Early Onset Anhydramnios Caused by Renal Anomalies: Background and Rationale for the Renal Anhydramnios Fetal Therapy Trial. Fetal Diagn Ther. 2019;45(6):365-372. doi: 10.1159/000497472. Epub 2019 Mar 21. PMID 30897573
- See also: Renal Anhydramnios Fetal Therapy (RAFT) Trial Wesbite — https://raft-trial.org/
- See also: Fetal Care Center - Amnioinfusion FAQ — https://fetalcaredallas.com/blog/what-is-amnioinfusion/